CLINICAL TRIAL: NCT02652117
Title: Retrospective Review of Regional Anesthesia in Cardiac Pediatric Patients
Brief Title: Regional Anesthesia in Cardiac Pediatric Patients Less Than 5 Years Old
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Other Study IDs: 201212725
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This retrospective review presents a comparison of pediatric patients less than 5 years old undergoing cardiac surgery with general anesthesia with spinal, caudal epidural, or caudal epidural with catheter anesthesia from July 2007 to July 2013 observing differences in time to extubation, reintubation, and hypercarbia.

DETAILED DESCRIPTION:
Intra-operative anesthesia medical records of pediatric patients undergoing cardiac surgery will be acquired from July 2007 to July 2013. Allocation of regional anesthesia, and the use of spinal versus epidural versus epidural with catheter administration will be determined by provider preference. Date of surgery, age in months, gender, type of surgery, type of anesthesia, regional drugs, PaCO2 upon arrival in the PICU, time to extubation, and reintubation if applicable will be recorded. Time to extubation will be categorized into within the OR, less than 24 hours, or greater than or equal to 24 hours. PaCO2 levels will be categorized into hypercarbia (PaCO2 ≥ 50mmHg) and normal (PaCO2 < 50mmHg).

ELIGIBILITY:
Inclusion Criteria:

* Must be pediatric patients undergoing cardiac surgery under the age of 5 years old between the years 2007 and 2013

Exclusion Criteria:

* None

Max Age: 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cardiac Pediatric Patients less than 5 years old
Sampling Method: Non-Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2007-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To expect difference in time to extubation | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sudhakar Subramani, MD, Principal Investigator — University of Iowa

REFERENCES:
- [Background] Fawcett WJ, Edwards RE, Quinn AC, MacDonald IA, Hall GM. Thoracic epidural analgesia started after cardiopulmonary bypass. Adrenergic, cardiovascular and respiratory sequelae. Anaesthesia. 1997 Apr;52(4):294-9. doi: 10.1111/j.1365-2044.1997.80-az0088.x. PMID 9135178
- [Background] Liu S, Carpenter RL, Neal JM. Epidural anesthesia and analgesia. Their role in postoperative outcome. Anesthesiology. 1995 Jun;82(6):1474-506. doi: 10.1097/00000542-199506000-00019. No abstract available. PMID 7793661